CLINICAL TRIAL: NCT02496000
Title: Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Multiple Oral Bedtime Doses of ORMD-0801 in Adult Patients With Type 2 Diabetes Mellitus Who Are Inadequately Controlled With Diet and Metformin
Brief Title: Phase II Safety and Efficacy Study of Oral ORMD-0801 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-007
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Type 2
Keywords: Diabetes Mellitus type 2; Metformin; oral insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ORMD-0801; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo Comparator (Placebo Comparator): three identical capsules containing placebo
  Interventions: Drug: Placebo Comparator
- ORMD-0801 Dose 1 (Experimental): three identical capsules, as follows: capsule #1: one half of Dose 1 capsule #2: one half of Dose 1 capsule #3: placebo
  Interventions: Drug: ORMD-0801
- ORMD-0801 Dose 2 = 1.5 * Dose 1 (Experimental): three identical capsules, as follows: capsule #1, 2, and 3: one half of Dose 1
  Interventions: Drug: ORMD-0801

INTERVENTIONS:
Drug: ORMD-0801 — Oral Insulin
  Other Names: Oral Insulin
  Arms: ORMD-0801 Dose 1; ORMD-0801 Dose 2 = 1.5 * Dose 1
Drug: Placebo Comparator — Placebo
  Other Names: Placebo
  Arms: Placebo Comparator

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel group study.

DETAILED DESCRIPTION:
This is a multicenter, Phase II, randomized, double-blind, placebo-controlled, parallel group study. After appropriate screening, approximately 180 male and female patients from up to 33 study centers will be treated in this study. Patients with type 2 diabetes mellitus who are being treated by diet, exercise, untreated with antidiabetic medications or treated with and metformin monotherapy or in combination with one other antidiabetic drug (excluding insulin) are eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c ≥7.5% if naïve to antidiabetic therapy; ≥6.5% and ≤10% if on metformin ≥1,500 mg daily; ≥6.5% and ≤9.5% if on monotherapy with an antidiabetic drug other than metformin; ≥ 6.5% and ≤9.5% if on metformin and one other antidiabetic drug; ≥ 7.0% if on metformin <1,500 mg daily.
* At time of randomization, patients will be treated for their diabetes by diet, exercise, and metformin (≥1500 mg/day; any type and regimen). Patients will have been on a stable regimen of metformin (defined as the same metformin dose and type) for at least two weeks prior to entering the single-blind placebo run-in period.
* Other antidiabetic agents will not be used for the two weeks prior to entering the placebo run-in period.
* Patients in whom the maximum tolerated dose (MTD) of metformin is 1,000 mg will be allowed to enter the study.
* At Day -7 (Visit 3), all patients will have HbA1c ≥ 6.5% and ≤10%.
* Body Mass Index between 25 and 40 kg/m2, inclusive.
* Fasting blood glucose ≥ 126 mg/dL (8.3 mmol/L) prior to randomization at Day -7 (Visit 3). For patients in whom the Day -7 (Visit 3) fasting blood glucose is <126 mg/dL and ≥ 115 mg/dL, and the Day -7 (Visit 3) HbA1C is ≥ 7% and ≤ 10%, a minimum of 5 daily self- monitored fasting blood glucose checks recorded in the patient diary can be averaged. If the average value is ≥ 126 mg/dL, the patient may continue in the trial.
* Females of childbearing potential must have a negative urine pregnancy test result at screening. A negative urine pregnancy test must be obtained during Visit 2 and at Visit 4 (prior to randomization).
* Males and females of childbearing potential must use two methods of contraception (double barrier method), one of which must be an acceptable barrier method from the time of screening to the last study visit (Day 43).
* Patient has >80% compliance with placebo during run in prior to randomization.
* Patient has ≥ 80% of the glucose readings on at least two 24 hour periods (6AM - 6AM) during the seven day CGM period.
* Patient has performed ≥ 10/14 of the self monitored glucose level measurements during placebo run-in, prior to randomization.

Exclusion Criteria:

- Patients who meet any of the following criteria are not eligible for this study.

* Presence of any clinically significant endocrine disease according to the Investigator (euthyroid patients on replacement therapy will be included if the dosage of thyroxine is stable for at least six weeks prior to Screening Visit).
* Clinical diagnosis of Type 1 diabetes.
* Fasting blood glucose >260 mg/dL at the end of Day -7/Visit 3. For patient in whom the Day 07 (Visit 3) fasting blood glucose is > 260 mg/dL and < 300 mg/dL, and the Day -7 (Visit 3) HbA1C is ≥ 7% and ≤ 10%, a minimum of 5 self-monitored fasting blood glucose checks recorded in the patient diary can be averaged. If the average value is ≤ 260 mg/dL, the patient may continue in the trial.
* Presence or history of cancer within the past five years with the exception of adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer.
* Laboratory abnormalities at screening including:

  1. C-peptide < 1.0 ng/mL.
  2. Positive pregnancy test in females of childbearing potential (at screening and start of run-in period).
  3. Abnormal serum thyrotropin (TSH) levels >1.5 times the upper limit of normal.
  4. Positive test for hepatitis B surface antigen and/or hepatitis C antibody.
  5. Positive test for HIV.
  6. Serum Cr >1.4mg/dl in males, >1.3mg/dl in females.
  7. Any relevant abnormality interfering with the efficacy or the safety assessments during study drug administration.
* Use of the following medications:

  1. History of use of insulin for greater than one week in the last six months and any use of insulin in the last six weeks prior to randomization.
  2. Administration of anti-diabetic drugs other than metformin within four weeks prior to randomization visit. Administration of thyroid preparations or thyroxine within six weeks prior to screening visit. (Patients on stable thyroid replacement therapy for greater than 6 weeks may enter the study.)
* Administration of systemic long-acting corticosteroids within two months or prolonged use (more than one week) of other systemic corticosteroids or inhaled corticosteroids within 30 days prior to screening visit.
* Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and inhaled steroids (as discussed above), beta blockers (with the exception of beta blocker ophthalmic solutions for glaucoma or ocular hypertension), and immunosuppressive or immunomodulating agents.
* History of tobacco or nicotine use in excess of two packs/day within ten weeks prior to screening.
* Patient is on a weight loss program and is not in the maintenance phase, or patient that started any approved or non approved weight loss medication within eight weeks prior to screening.
* Pregnancy or breast-feeding.
* Patient has a screening visit systolic blood pressure of ≥160 mm Hg or diastolic blood pressure of ≥100 mm Hg Patients will be allowed to take BP medication as long as they have been on a stable dose for a period of four weeks prior to the screening visit.
* Patient is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week, or binge drinking).
* Elevated liver enzymes (alanine transaminase (ALT), alanine aminotransferase (AST), alkaline phosphatase) greater than two times the upper limit of normal at screening.
* Very high triglyceride level (>500 mg/dL) at screening.
* Any clinically significant electrocardiogram (ECG) abnormality at screening or cardiovascular disease. Clinically significant cardiovascular disease will include:

  1. History of stroke, transient ischemic attack, or myocardial infarction within six months prior to screening,
  2. History of or currently have New York Heart Associate Class II-IV heart failure prior to screening, or
  3. Uncontrolled hypertension defined as blood pressure ≥160 mmHg (systolic) or ≥100 mmHg (diastolic) at screening.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, M.D., Principal Investigator — Orange County Research Center
Locations (34):
- United States (34):
  - Steingard Medical Group, Phoenix, Arizona
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - Dream Team Clinical Research, Anaheim, California
  - ACTCA, Inc., Los Angeles, California
  - ACTCA, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Providence Clinical Research, North Hollywood, California
  - Mills-Peninsula Health Services, San Mateo, California
  - Orange County Research Center, Tustin, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Research in Miami Inc., Hialeah, Florida
  - Research in Miami, Inc., Hialeah, Florida
  - Phoenix Medical Research LLC, Miami, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Metabolic Research Institute, Inc, West Palm Beach, Florida
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Maine Research Associates, Auburn, Maine
  - Apex Medical Research, MI, Inc, Flint, Michigan
  - Impact Clinical Trials, Las Vegas, Nevada
  - New York Clinical Trials, New York, New York
  - Lynn Institute of Norman, Norman, Oklahoma
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Padre Coast Clinical Research, Corpus Christi, Texas
  - Sun Research Institute, San Antonio, Texas
  - Southwest Clinic, San Antonio, Texas
  - Panacea Clinical Research, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Rainier Clinical Research Center, Inc., Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study design: screening, followed by a 14 day wash-out followed by a 14-day single-blind run-in prior to the 28-day treatment period. Efficacy based on the Intend-to-treat population 80% trimming of the data. The safety (adverse events) data is based on the safety population.
Period: Overall Study
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1
Started | 64 | 61 | 63
Completed | 62 | 56 | 61
Not Completed | 2 | 5 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Non-compliance or lack of cooperation | 0 | 2 | 0
Not completed — undetermined | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1 | Total
Number analyzed (Participants) | 64 | 61 | 63 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.61 (9.203) | 57.89 (8.021) | 57.25 (8.786) | 57.92 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 22 | 29 | 86
  Male | 29 | 39 | 34 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 32 | 36 | 99
  Not Hispanic or Latino | 33 | 29 | 27 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 7 | 8 | 4 | 19
  White | 53 | 50 | 55 | 158
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Measure of the Mean Night Time Glucose Levels Based on Two Nights of Glucose Measurements.
Description: The Effect of ORMD-0801 (Doses 1 & 2, Pooled) on Mean Night Time Glucose Levels (measured in mg/dL) Based on 2 Nights of Continuous Glucose Monitor (CGM) Data by Comparison of the Mean Change Between Baseline and Wk 4 of ORMD-0801 Treatment and Placebo Groups. The primary analysis will be based on the results from the two last days, unless technical difficulties preclude calculation of the weighted mean glucose levels. In this case, the last two days (selected between days 5, 6, and 7) with at least 80% of the expected number of measurements will be used. If days 5, 6 and 7 do not have 2 days with at least 80% of the expected number of measurements for a specific subject, then the value will be missing for that subject.
Time Frame: Baseline-Study day -7 (± 1 day) through Study day 1 (± 1 day), and Week 4 -Study day 22 (± 1 day) through Study day 29 (± 1 day)
Population: Intend-to-Treat Population, 80% trimming. The mean values will be analyzed using a one-way analysis of variance (ANOVA) model. The residuals from the ANOVA will be analyzed to verify that they are normally distributed. If not normally distributed, then a Kruskal-Wallis test (one-way analysis of variance on the ranks) will be performed.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- ORMD-0801 Doses 1 and 2 Combined: The combined measurements of dose 1 and dose 2, in units of mg/dL
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1 | ORMD-0801 Doses 1 and 2 Combined
Number analyzed (Participants) | 46 | 44 | 47 | 91
mg/dL | 13.70 (26.140) | -3.67 (18.983) | 6.64 (26.361) | 1.66 (23.541)
Statistical Analysis 1: Comparison: Placebo Comparator vs ORMD-0801 Dose 1 vs ORMD-0801 Dose 2 = 1.5 * Dose 1; This outcome measure requires that the the mean differences of ORMD-0801 in each of the two arms be pooled; Test type: Superiority or Other; p = 0.0117, Kruskal-Wallis; ANOVA model on the ranks

2. Secondary Outcome: The Effect of ORMD-0801 on Mean 24-hour Glucose
Description: The effect of ORMD-0801 (Dose 1 and Dose 2 individually) on mean 24-hour glucose based on 2 nights of CGM data by comparison of the mean percent change between baseline and Wk 4 of ORMD-0801 treatment and the placebo groups.
Time Frame: Study day -7 (± 1 day) through Study day 1 (± 1 day), and Study day 22 (±1 day) - Study day 29 (± 1 day)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1
Number analyzed (Participants) | 56 | 54 | 59
percent change | 5.34 (13.881) | 3.33 (21.499) | 1.93 (19.795)

3. Secondary Outcome: Measure Percent Change in Continuous Glucose Monitoring Mean Fasting Glucose Between Treatment and Run-In
Description: The percent change in the Continuous Glucose Monitoring Mean Fasting Glucose between treatment and mean of the last two days of the baseline(run-in period).
Time Frame: Baseline (Run-in days 13-14) and Study day 1 (± 1 day) through Study day 29 (± 1 day)
Population: Intend to Treat (ITT)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1
Number analyzed (Participants) | 58 | 54 | 58
percent change | 12.76 (23.245) | 4.54 (24.153) | 3.28 (27.331)

4. Secondary Outcome: Measure the Change From Baseline to End of the Study of Morning Fasting C-Peptide (Nmol/L)
Description: The measurement of the change in Morning Fasting C-peptide between baseline to end of the study, measured in Nmol/L
Time Frame: Study day 1 (±1 day) through Study day43 (± 1 day)
Population: Intend to Treat (ITT) population
Measure: Mean (Standard Deviation); unit: Nmol/L
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1
Number analyzed (Participants) | 54 | 54 | 58
Nmol/L | 0.08 (0.252) | 0.03 (0.476) | 0.7 (0.300)

5. Secondary Outcome: The Effect of ORMD-0801 on the Percent Change in HbA1c
Description: The effect of ORMD-0801 (Dose 1 and Dose 2 individually) on the percent change from baseline to Wk 4 in HbA1c
Time Frame: Study day 1 (± 1 day) through Study day 29 (± 1 day)
Population: Intend To Treat (ITT) population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1
Number analyzed (Participants) | 58 | 53 | 59
percent change | 0.2 (0.497) | 0.00 (0.544) | -.03 (0.554)

ADVERSE EVENTS:
Time Frame: eight (8) months
Arm/Group | Placebo Comparator | ORMD-0801 Dose 1 | ORMD-0801 Dose 2 = 1.5 * Dose 1
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/61 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/61 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator (N=64) | ORMD-0801 Dose 1 (N=61) | ORMD-0801 Dose 2 = 1.5 * Dose 1 (N=63)
Serious Non-Treatment Emergent Adverse Event (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Basal Ganglia Stroke

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days